CLINICAL TRIAL: NCT00742157
Title: An Open-label Evaluation of the Long-term Efficacy and Safety of a Standardized Regimen of Growth Hormone, Glutamine and a Modified Diet in the Treatment of Patients With Short Bowel Syndrome
Brief Title: Evaluate the Efficacy and Safety Growth Hormone, Glutamine and Diet in Patients With Short Bowel Syndrome (SBS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: University of Nebraska (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0061-03-FB
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Results first posted 2023-07-28 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Short Bowel Syndrome
Keywords: Growth Hormone; TPN; Total Parenteral Nutrition; Glutamine; Short Bowel Syndrome; Increase in absorption of small bowel.
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — Growth Hormone; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UNMC Group (Other): Compare the low and high dose effects of Growth Hormone from previously pooled patients (high dose) and UNMC patients (low dose).
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — dosage = 0.05mg/kg/day, in diluent for injection, once a day, for 23 - 54 days.
  Other Names: Humatrope = Somatropin (rDNA origin) for injection

SUMMARY:
Treatment for 3.5-8 weeks with GH (0.05 mg/kg/day) +GLN+Diet, followed by continued compliance to the individualized oral diet and enteral GLN, will result in reduced volume of TPN infusion/week and/or reduced frequency of TPN infusions/week.

DETAILED DESCRIPTION:
Long-term total parenteral nutrition (TPN) is a supportive, rather than curative, therapy for patients with severe short bowel syndrome (SBS). Because of the complications (liver and kidney dysfunction, bone demineralization, nutrient deficiencies, catheter sepsis) and costs (>$100,000/ patient/year) associated with this therapy, researchers have attempted to identify a safe, cost-effective alternative treatment modality. Various surgical procedures (including bowel transplantation) have been explored; however, these options currently offer limited clinical efficacy and significant morbidity and mortality. In contrast, a non-invasive therapy utilizing a growth factor (growth hormone - GH) and a bowel-specific nutrient (glutamine - GLN) in combination with an individualized oral diet (GH+GLN+Diet) has recently been shown to significantly enhance nutrient absorption and eliminate or reduce TPN requirements in patients with severe SBS.

This open-labeled, single-center trial with a total enrollment of 30 patients with severe SBS will examine the safety and effectiveness of a lower dose (0.05 mg/kg/day) of growth hormone. Thirty-two subjects have previously been studied at the Nutritional Restart Center in Massachusetts utilizing a higher dose (0.1 mg/kg/day) of growth hormone and identical treatment parameters as described in this protocol. The University of Nebraska Medical Center and the Nutritional Restart Center have agreed to pool the data from both studies and analyze the data according to the same primary efficacy variable. Subjects recruited to the lower-dose growth hormone group will be matched, using specific clinical criteria, to patients in the higher dose growth hormone group. The primary efficacy variable will be the change in volume of TPN infusion/week and frequency of TPN infusions/week at 6 months following discharge compared to baseline.

After a 3 day, baseline evaluation at The Nebraska Medical Center to determine pre-treatment TPN requirements and to assess the specific indices of nutritional and hydration status and kidney and liver function, and physical functioning capacity, patients will begin to receive lower dose GH (0.05 mg/kg/day) in combination with GLN (30 grams/day, orally) and the individualized oral/enteral diet. Treatment will last for a minimum of 23 days and a maximum of 54 days. Duration of treatment will be tailored to the patients' individual needs (e.g., understanding and acceptance of the modified diet, successful weaning of TPN). Patients may return to their home to continue receiving the GH treatment, provided they are tolerating the GH injections and understand how to properly administer the injections.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between 19 and 78 years of age, inclusive
* Have a diagnosis of SBS and 1 or more of the following characteristics:
* Dependent upon TPN and/or IV fluids
* Unable to receive TPN because of a documented history of complications associated with the long-term parenteral infusions (e.g. lack of venous access, multiple septic events, progressive liver dysfunction while on TPN, etc)
* A documented remnant bowel anatomy that is inconsistent with adequately supporting life without parenteral support (e.g. < 70 cm of healthy small intestine and a portion of colon, or less than 150 cm in patients with no colon)
* A documented history of diarrhea and/or malabsorption that has significantly compromised the patient's nutritional and hydration status (e.g. significant weight loss - 5% over 1 month or 10% over 6 months, or a serum albumin < 3.5 g/dl, documented nutrient deficiencies, documented episodes of dehydration, etc).
* Is able to eat at least some (>500 calories) of solid food on a regular basis or tolerate at least some (>500 calories) of an enteral feeding formula
* Have stable liver and renal function
* For patients with known hypertension and other cardiovascular disorders, be both compensated and stabilized on a regular therapeutic regimen
* For women participating in the study, manifest or give assent to 1 of the following criteria to ensure that the patient does not become pregnant during the study:
* The patient must be surgically sterile or demonstrably postmenopausal.
* Any patient capable of becoming pregnant must have a negative urine pregnancy test and must agree to practice a method of contraception documented to have at least 90% reliability throughout the treatment period.
* Have the ability to understand the requirements of the study, to provide written Informed Consent, and to abide by the study restrictions and agree to complete the required assessments in the Follow-up Period

Exclusion Criteria:

* Be pregnant or lactating
* Have a history of mental deficiency or illness that might compromise compliance with the requirements of the study
* Have clinically serious neurological dysfunction
* Have hypoxemic pulmonary diseases (i.e., resting pAO2 < 75 torr)
* Have unstable ischemic heart disease or uncompensated cardiac failure
* Have participated in any study involving an investigations drug within 30 days prior to entry into this trial.

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2008-10-20 (Actual); Study Completion 2008-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fedja Rochling, MB, ChB, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (n=5) were recruited between 9/2003 and 4/2008 in a gastroenterology clinic in the university hospital ( single site)
Groups:
- Single Arm Protocol: An Open-label Evaluation of the Long-term Efficacy and Safety of a Standardized Regimen of Growth Hormone, Glutamine and a Modified Diet in the Treatment of Patients with Short Bowel Syndrome
Period: Overall Study
Arm/Group | Single Arm Protocol
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.6 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Documenting the Reduction of TPN Infusion/Week for Participants at 6 Months Compared to Baseline.
Description: Evaluate the number of participants dosed at UNMC who had a reduction in the frequency of TPN infusions/week at 6 months compared to baseline
Time Frame: 6 months
Population: 5/5 participants dosed at UNMC had a reduction in the frequency of TPN infusions/week at 6 months compared to baseline.
Measure: Count of Participants; unit: Participants
Groups:
- UNMC Group: Participants dosed at UNMC with 0.05mg/kg/day in diluent for injection, once a day for 23-54 days
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Change in Hydration Status
Description: Number of participants who were able to maintain euvolemic status at 6 months post treatment
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
participants | 5

3. Secondary Outcome: Change in Kidney Function at 6 Months Post Treatment
Description: Number of participants with a significant change in kidney function at 6 months post treatment as compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Change in Liver Function at 6 Months Post Treatment
Description: Number of participants with an improvement in their liver function ALT at 6 months post treatment as compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
Participants | 2

5. Secondary Outcome: Change in Physical Functioning Capacity at 6 Months Post Treatment as Compared to Baseline
Description: Number of participants who had a change in their ability to complete all activities of daily living by self at 6 months compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | UNMC Group
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- UNMC Group: Group of subjects (n=5) who received treatment
Arm/Group | UNMC Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UNMC Group (N=5)
bacteremia (Infections and infestations) | 1 (1) — staphylococcus epidermidis line infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UNMC Group (N=5)
edema (Cardiac disorders) | 1 (1) — bilateral ankle edema
hyperglycemia (Endocrine disorders) | 1 (1) — hyperglycemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes